CLINICAL TRIAL: NCT02993666
Title: Comparison of Upper and Lower Body Air Warming in Patients Undergoing Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong-Hwa Seo, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JHSeo_FAW
Record Dates: First submitted 2016-12-01; First posted 2016-12-15 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Core Body Temperature

ARMS (2):
- upper body (Experimental): warming with upper body blankets
  Interventions: Device: Bair Hugger
- lower body (Experimental): warming with lower body blankets
  Interventions: Device: Bair Hugger

INTERVENTIONS:
Device: Bair Hugger — forced air warming with Bair Hugger air warmer

SUMMARY:
This study is conducted to evaluate the effectiveness of forced air warming using upper and lower body blankets by measuring core body temperature in patients undergoing video-assisted thoracic surgery in the lateral decubitus position over 2 hours of general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing video-assisted thoracic surgery over 2 hours
* ASA I, II and III
* age over 18 years

Exclusion Criteria:

* refuse to enroll
* patients with fever or hypothermia before surgery
* patients who required changes of position during surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
intraoperative incidence of hypothermia | through surgery completion, up to 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: JH Seo, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Min SH, Yoon S, Yoon SH, Bahk JH, Seo JH. Randomised trial comparing forced-air warming to the upper or lower body to prevent hypothermia during thoracoscopic surgery in the lateral decubitus position. Br J Anaesth. 2018 Mar;120(3):555-562. doi: 10.1016/j.bja.2017.11.091. Epub 2017 Dec 5. PMID 29452812